CLINICAL TRIAL: NCT02063958
Title: A Phase 1, Open-label, Dose-escalation Study of SNX 5422 and Everolimus in Subjects With Neuroendocrine Tumors.
Brief Title: Safety and Pharmacology of SNX-5422 Plus Everolimus in Subjects With Neuroendocrine Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Esanex Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SNX5422-CLN-009
Record Dates: First submitted 2014-02-13; First posted 2014-02-17 (Estimated); Last update posted 2018-07-30 (Actual); Status verified 2018-07

CONDITIONS: Cancer
Keywords: Neuroendocrine tumor; Hsp90
MeSH Terms: conditions — Neoplasms; Neuroendocrine Tumors | interventions — SNX-5422

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SNX-5422 (Experimental): Open-label administration of SNX-5422 capsules dosed in the morning once every other day (qod) for 21 days (11 doses), followed by a 7 day drug free period. Dose escalation will be based on safety defined as 1 or less dose limiting toxicities during the first 28 day cycle at any dose level. Dose escalation will not exceed a dose of 100 mg/m2 SNX-5422 qod even if the MTD has not been identified. Subjects will receive daily oral everolimus in the PM about the same time every day for 28 days.
  Interventions: Drug: SNX-5422

INTERVENTIONS:
Drug: SNX-5422 — Capsule dosed every other day for 21 days out of a 28 day cycle. Dose escalation based on safety not to exceed a dose of 100 mg/m2. Maintenance therapy of SNX-5422 at the MTD will be allowed for all patients not experiencing significant toxicity.

SUMMARY:
Study is designed to determine the maximum tolerated dose (MTD) of SNX-5422 when given in combination with everolimus.

DETAILED DESCRIPTION:
Heat shock protein 90 (Hsp90) plays a central role in the maturation and maintenance of numerous proteins, for example HER2 and mutated EGFR, that are critical for tumor cell viability and growth; SNX-5422 is a pro-drug of SNX-2112, a potent, highly selective, small-molecule inhibitor of the molecular chaperone heat shock protein 90 (Hsp90). Hsp90 has been found to be expressed in 95% of subjects with pancreatic neuroendocrine tumors.

This study will determine the MTD of SNX-5422 when given in combination with everolimus in patients with neuroendocrine tumors.The clinical starting dose of 50 mg/m2 qod for SNX-5422 in combination with daily everolimus is 50% of the SNX-5422 qod mono-therapy MTD. The choice to continue once every other day SNX-5422 dosing is based on the safety and efficacy profiles from prior studies, so that drug holidays are interspersed into weekly dosing. The planned subsequent dose levels are 75% and 100% of the SNX-5422 qod mono-therapy MTD.

ELIGIBILITY:
Inclusion Criteria:

* Males or non-pregnant, non-breastfeeding females 18 years-of-age or older.
* Archived neuroendocrine tumor sample or biopsy sample (will also be used for genetic testing).
* Pathologic evidence of chemo-resistant Small Cell Lung cancer (relapse <90 days after 1st line), chemo-sensitive Small Cell Lung Cancer (relapse >90 days after first line), locally advanced metastatic neuroendocrine tumor of gastro-entero, pancreatic, pulmonary (other than Small Cell Lung) or thymic origin, or advanced renal cell carcinoma for which everolimus is indicated.
* Measurable (RECIST) indicator lesion not previously irradiated.
* Life expectancy of at least 3 months.
* No more than 4 prior lines of systemic anti-cancer therapy.
* Karnofsky performance score ≥70.
* Adequate baseline laboratory assessments, including

  * Absolute neutrophil count (ANC) ≥1.5 x 109/L.
  * WBC >3000/microliter
  * Platelet count of ≥100 x 109/L.
  * Total bilirubin level ≤1.5 times institutional upper limit of normal (ULN), alanine aminotransferase or aspartate aminotransferase ≤2 x ULN
  * Hemoglobin ≥9 mg/dL.
  * Creatinine <1.5 X upper limit of normal or estimated plasma creatinine clearance of ≥40 mL/min
* Signed informed consent form
* Recovered from toxicities of previous anticancer therapy
* Subjects with reproductive capability must agree to practice adequate contraception methods.

Exclusion Criteria:

* Subjects in whom everolimus is contraindicated.
* Subjects with clinically significant interstitial lung disease, or obstructive disease without sufficient reserve
* Carcinoid with hormone related symptoms
* Neuroendocrine cancer of the thyroid or thymus.
* Rare pancreatic neuroendocrine cancers such as, insulinomas, glucagonomas, gastrinomas.
* Prior treatment with any Hsp90 inhibitor.
* Prior failed treatment with mTOR inhibitors
* CNS metastases that are symptomatic and /or requiring escalating doses of steroids.
* Major surgery or significant traumatic injury within 4 weeks of starting study treatment.
* Conventional chemotherapy or radiation within 4 weeks.
* Palliative radiation within 2 weeks.
* The need for treatment with medications with clinically-relevant metabolism by the cytochrome P450 (CYP) 3A4 isoenzyme within 3 hours before or after administration of SNX-5422
* Screening ECG QTc interval ≥470 msec for females, ≥450 msec for males.
* At increased risk for developing prolonged QT interval, including hypokalemia or hypomagnesemia, unless corrected to within normal limits prior to first dose of SNX-5422; congenital long QT syndrome or a history of torsade de pointes; currently receiving anti-arrhythmics or other medications that may be associated with QT prolongation.
* Patients with chronic diarrhea or with Grade 2 or greater diarrhea despite appropriate medical management.
* Gastrointestinal diseases or conditions that could affect drug absorption, including gastric bypass.
* Gastrointestinal diseases that could alter the assessment of safety, including irritable bowel syndrome, ulcerative colitis, Crohn's disease, or hemorrhagic coloproctitis.
* History of documented adrenal dysfunction not due to malignancy.
* Known seropositive for human immunodeficiency virus (HIV) or hepatitis C virus (HCV).
* History of chronic liver disease.
* Active hepatitis A or B.
* Current alcohol dependence or drug abuse.
* Use of an investigational treatment from 30 days prior to the first dose of SNX-5422 and during the study.
* Glaucoma, retinitis pigmentosa, macular degeneration, or any retinal changes detected by ophthalmological examination.
* Other serious concurrent illness or medical condition.
* Psychological, social, familial, or geographical reasons that would hinder or prevent compliance with the requirements of the protocol or compromise the informed consent process.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2017-03-27 (Actual); Study Completion 2018-03-20 (Actual)

PRIMARY OUTCOMES:
Number of patients with dose limiting toxicities | First 28 day cycle
  Number of patients with dose limiting toxicities defined as adverse events or laboratory abnormalities of Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 ≥ Grade 3 that are not clearly related to disease progression or delay by more than 4 weeks in receiving the next scheduled cycle due to persisting toxicities and attributable to the combination of SNX-5422 and everolimus despite optimal medical supportive management.

SECONDARY OUTCOMES:
Number of patients with adverse events as a measure of tolerability | Every 4 weeks
  Frequency and severity of adverse events
Changes in ECG, vital signs, laboratory or physical examination | Every 4 weeks
  Changes in ECG, vital signs, laboratory or physical examination from baseline
Tumor response | Every 8 weeks
  Measurements from tumor imaging within 1 month prior to the screening visit will be used as the baseline assessment. This assessment will be performed using Response Evaluation Criteria in Solid Tumors (RECIST 1.1). Follow-up imaging of known sites of the disease, preferably by CT scan, will be performed at intervals appropriate to the subject's disease and clinical findings.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Mayo Clinic, Scottsdale, Arizona
  - Stanford Medicine, Stanford, California
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Center for Cancer Research, National Cancer Institute, Bethesda, Maryland
  - hackensack University Medical Center, Hackensack, New Jersey